CLINICAL TRIAL: NCT04893616
Title: Improving Timeliness of Birth Dose Vaccines in 15 Health Facilities in Cameroon Through Integrating Immunizations Into Maternity and Newborn Care Services: A Feasibility Assessment
Brief Title: Cameroon HepB Birth Dose Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Cameroon Expanded Program on Immunization (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/09/1695/L/CNERSH/SP
Record Dates: First submitted 2021-03-17; First posted 2021-05-19 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): These facilities will be those selected to have the intervention carried out.
  Interventions: Other: Integration of vaccination services into delivery services

INTERVENTIONS:
Other: Integration of vaccination services into delivery services — The purpose of the work is to integrate readily available birth dose vaccinations (Oral Polio and the Tuberculosis vaccine) currently given in a separate clinic into the maternity delivery services through improved training, checklist, and job aides.

SUMMARY:
This feasibility assessment is to provide quantitative findings of an intervention integrating immunizations into maternity and newborn care across 15 health facilities in Cameroon.

DETAILED DESCRIPTION:
In the Cameroon Expanded Program on Immunization (EPI), the birth dose vaccine for oral polio vaccine (OPV-0) and tuberculosis vaccine (BCG), are recommended with a third birth dose vaccine for hepatitis B (HepB-BD) being considered for introduction.

Although Cameroon introduced the HepB antigen as part of the Pentavalent vaccine into the immunization program in 2005, infants are currently unprotected until the first Penta shot at six weeks. Introduction of HepB-BD is a key priority for the Cameroon government through the National Cancer Strategy document as well as the Hepatitis Prevention and Treatment Guidelines. However, the timeliness of administration of Hepatitis B vaccine within 24 hours of birth is critical to ensure the highest efficacy and prevent transmission of the virus.

While coverage rates for BCG and OPV 0 are relatively high (91% and 78% respectively), these vaccines are often administered weeks or months after birth , not within the 24-hour timeframe recommended for Hepatitis B birth dose. Therefore, there are concerns from the Cameroon National Immunization Technical Advisory Group (NITAG) and other stakeholders on the feasibility of achieving high timely coverage of HepB-BD. The timeliness of administration of the birth dose vaccines within facilities relies on many system components including integrated processes between maternity and immunization units and healthcare worker awareness of birth dose administration guidelines.

The main aim of this pilot study is to assess the feasibility of immunizing newborns with BCG and OPV0 (and eventually HepB-BD) within 24 hours of birth by integrating routine immunization into maternity and immediate newborn care in 15 facilities in Cameroon.

Further, the specific objectives of this pilot study are to:

1. Integrate birth dose immunizations into maternity and immediate newborn care services
2. Measure the change in proportion of newborn receiving birth doses BCG and OPV0 within 24 hours compared to baseline data
3. Measure the change in average age of babies receiving birth doses of BCG and OPV0
4. Assess the operational feasibility and acceptability of interventions and describe any factors (barriers and enablers) that may influence further implementation of birth dose strategies

This feasibility assessment is to provide quantitative findings of an intervention integrating immunizations into maternity and newborn care across 15 health facilities in Cameroon. Overall, in 20 weeks an intervention phase will be followed by a final assessment. The approach will utilize quantitative data from healthcare worker surveys, the birth registry and immunization registry, and maternity unit reporting forms. The study findings will be used to inform strategy on HepB-BD introduction in Cameroon as well as interventions to strengthen service delivery structures for newborns.

ELIGIBILITY:
Inclusion Criteria:

* Facilities will be those that have both an immunization unit as well as a maternity ward

Exclusion Criteria:

* Facilities without both units

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Timeliness of birth dose vaccine administration | 20 weeks
  Median hours between birth and administration of oral polio and/or the BCG vaccine

SECONDARY OUTCOMES:
Coverage of birth dose vaccines | 20 weeks
  The proportion of children born in the facility that obtain an oral polio and/or BCV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Ankouane Andoulo Firmin, Principal Investigator — Faculty of Medicine and Bio-Medical Sciences, University of Yaoundé
Locations (13):
- Cameroon (13):
  - CMA Dibi, Dibi, Adamaoua Region
  - CMA Mbe, Mbé, Adamawe
  - HD Biyem-Assi, Biyem Assi, Center
  - HD Cite Verte, Cite Verte, Center
  - CMMR Etoudi, Djoungolo, Center
  - CMA Ahala, Efoulan, Center
  - CSIU Mbalmayo II, Mbalmayo, Center
  - CSC Nkoabang, Mfou, Center
  - Hospital Nicolas Barre, Nkolndongo, Center
  - HD Obala, Obala, Center
  - CSC Baham, Baham, West Region
  - HD Foumbot, Foumbot, West Region
  - HD Mifi, Mifi, West Region

IPD SHARING:
Plan to Share IPD: No
Data on individual participant data will not be shared with other researchers. All reports will have data aggregated to the facility level. No personal identifiers will be gathered.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT04893616/Prot_SAP_ICF_000.pdf